CLINICAL TRIAL: NCT06375889
Title: Platelet Activation in Delayed Cerebral Ischemia Secondary to Aneurysmal Subarachnoid Hemorrhage
Acronym: APICRASH
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0250; 2024-A00796-41 (Other: ID-RCB)
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Aneuvrysmal Subarachnoid Hemorrhage; Delayed Cerebral Ischemia; Endotheliopathy; Platelets Kinetic
Keywords: aSHA; DCI; Endotheliopathy; Platelets
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2,7mL blood sample at day 0, 3, 5, 7, 10 (Total = 13,5mL) No other specimen required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- aSAH group: Patient hospitalised following the occurrence of an aneurysmal subarachnoid haemorrhage of any grade of severity.
  Interventions: Other: blood test
- IPH group: Patient hospitalised following the occurrence of a non-traumatic intra-parenchymal haematoma.
  Interventions: Other: blood test

INTERVENTIONS:
Other: blood test — During the routine blood test of the patient, 5 more tubes of 2.7 milliliters (mL) will be collected to make Platelet Activation Analysis

SUMMARY:
Aneurysmal subarachnoid haemorrhage is a complex pathology, the pathophysiology of which is still imperfectly understood. Its morbidity and mortality remain significant. In addition to the damage sustained by the brain in the immediate aftermath of aneurysmal rupture, which is inaccessible to life-saving treatment, a significant proportion of lesions occur at a distance from the initial event. Delayed cerebral ischaemia is one of the most morbid complications. It combines an inflammatory pattern with vascular dysfunction and neuronal excitotoxicity, leading to avoidable secondary neuronal loss.

Vascular dysfunction is mediated by a loss of homeostasis between endothelial cells and figurative blood cells, including platelets. However, the interrelationship between these elements and the precise chronology of the dysfunction remain imperfectly described to date.

It therefore seems appropriate to propose temporal monitoring of platelet activation kinetics over time, combined with concomitant collection of markers of endothelial damage, in order to clarify the vascular chronobiology of this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Adults ≤18 years of age.
* Hospitalised in the neurological intensive care unit of the Pierre Wertheimer Hospital of the Hospices Civils de Lyon following an aneurysmal meningeal haemorrhage of any modified Fischer score, previously diagnosed by cerebral CT scan.
* Patients admitted to the neurological intensive care unit or the NICU of the Pierre Wertheimer Hospital of the Hospices Civils de Lyon for an intra-parenchymal haematoma.
* Patient who has been informed and has formulated his/her non-opposition, or close relative of the patient who has been informed and has formulated his/her non-opposition.
* Affiliated to a social security scheme.

Exclusion Criteria:

* Non-aneurysmal SAH
* Ischaemic stroke
* Patients with previously known platelet function disorders
* Pregnant or breast-feeding women
* Patients under legal protection (guardianship, curatorship, safeguard of justice)
* Patients under compulsory psychiatric care
* Patients taking part in a study which may interfere with the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We therefore chose to carry out an exhaustive recruitment of the active file of consecutive patients eligible for the study selection criteria. In the Medical ICA and Neurovascular ICU Department of the Pierre Wertheimer Hospital of the Hospices Civils de Lyon, treating patients with sub-aneurysmal meningeal haemorrhage or intraparenchymal haemorrhage. 40 patients in each group
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-01-24 (Actual); Study Completion 2026-01-24 (Actual)

PRIMARY OUTCOMES:
The difference in the percentage of platelets expressing P-selectin, reflecting their irreversible activation. | Day of blood sample (inclusion visit) Day 3, day 5, day 7 and day 10 after inclusion visit
  To describe the temporal kinetics of the percentage of activated platelets over time between patients with aHSA compared with the control group, consisting of patients with spontaneous intraparenchymal haematomas. Platelet cell activation is defined by the concomitant presence of the following markers: P-Selectin (CD-62); Gp Integrin Alpha IIb Beta 3 (CD-41); phosphatidylserine.
  A mixed effects linear regression model will be used for data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Chardon, MD;Msc, Principal Investigator — Intensive care department; Pierre Wertheimer Hospital
Locations (2):
- France (2):
  - Anaesthesiology and Intensive Care medicine department, Pierre Wertheimer hospital, Bron, Auvergne-Rhône-Alpes
  - Neurovascular intensive care unit department, Pierre Wertheimer hospital, Bron, Auvergnes-Rhones-Alpes